CLINICAL TRIAL: NCT04815629
Title: Outcome of Radical Radiation Therapy in Squampus Cell Carcinoma
Brief Title: Outcome of Radiation Therapy in Urinary Bladder Squampus Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Anter Ali, Principal investigator, Assiut University
Other Study IDs: Radiotherapy in bladder cancer
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Urinary Bladder Squamous Cell Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Radiotherapy — Radiotion therapy squamous cell carcinoma in cancer bladder

SUMMARY:
Detection of distribution of clinico-pathological features of squamous cell carcinoma of urinary bladder and their relation to treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 .
2. histologically proved urinary bladder squamous cell carcinoma.
3. non-metastatic disease.
4. all patients who underwent radical treatment or bladder preserving approach.
5. patient with isolated urinary bladder carcinoma (no other or previous primary).

Exclusion Criteria:

1. age < 18 , > 70.
2. patient not documented having bladder squamous cell carcinoma by biopsy (cystoscopic or operative).
3. metastatic disease.
4. patient with synchronous or metachronous double primary

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient with urinary bladder squamous cell carcinoma recieved radiotherapy .
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | baseline
  Disease free survival

REFERENCES:
- [Background] 1. Messing EM. Urothelial tumours of the bladder. In: Wein AJ, Kavoussi LR, Novick AC, Partn AW, Peters CA (editors). Campbell-Walsh Urology. 9th(3). Philadelphia: Saunders Elsevier 2007: pp.2407-2446. 2. Christopher Ho Chee Kong, Praveen Singam, Goh Eng Hong, Lee Boon Cheok, Muhammad Azrif, Azmi Mohd Tamil et.al (2010). Clinicopathological features of bladder tumours in a single insttuton in Malaysia. Asian Pasifc J cancer Prev. 2010; 11: 149-152. 3. Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ (2009). Cancer statstcs. CA Cancer J Clin. 2009 ; 59: 529-533. 4.Zarzour AH , Selim M, Abd -Elsayed A et al., muscle invasive bladder cancer in uppr Egypt : the shift in risk factors and tumor characteristics, license Bio Med central BMC Cancer doi.:10.1186 / 1471-2407-8-250-,2008. 5.Amal S. Ibrahim, Nabiel N Mikhail et al . Egypt National Cancer Registry Damietta profile - 2009: publication number RR2 July, 2011. 6.M.Nabil El- Bolkiny , M.Akram Nouh , Tarek N.El-Bolkiny et al.topographic pathology of cancer , the national cancer institute, Cairo University , 2008. 7.Jason A.Efstathiou, Anthony L.Zietman, Jhon J. Coen, clinical Radiation Oncology , bladder cancer ;3rd edition : p1216-1241, 2012.